CLINICAL TRIAL: NCT02365844
Title: Multispectral Imaging to Characterize Patterns of Vascular Supply Within the Lymphoepithelial Mucosa of Patients With Known or Suspected Oropharyngeal Carcinoma (OPC)
Brief Title: Multispectral Imaging to Characterize Patterns of Vascular Supply Within Lymphoepithelial Mucosa in Oropharyngeal Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: ENT0044
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Oropharyngeal Carcinoma; Oropharynx Cancer
Keywords: Narrow Band Imaging; oropharyngeal carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to characterize the blood supply at the base of the tongue and within the tonsil region. We hypothesize that high-resolution Narrow Band Imaging (NBI) will improve the diagnosis of oropharyngeal carcinoma (OPC). The goal is to provide the better assessment of tumor and thus providing better preoperative expectations to patients with OPC or tumor extent prior to radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* Written informed consent
* Patients with oropharyngeal carcinoma

Exclusion Criteria:

* Tumors of the oral cavity or nasopharynx

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stanford Cancer Center patients with oropharyngeal carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
assessment of differential vascularity between normal and clinically apparent tumor with in the specified sites of oropharynx, using standard white-light endoscopy and narrow-band imaging | 30 minutes
  endoscopy of the oropharynx using white-light and narrow-Band imaging

CONTACTS AND LOCATIONS:
Overall Officials: Chris Holsinger, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States